CLINICAL TRIAL: NCT06953544
Title: The Effect of Father-Sensitive Childbirth Education on Prenatal Paternal Attachment Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevil Güner (Other)
Responsible Party: Sponsor-Investigator, Sevil Güner, Assistant Professor, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MERSINU*GHOSHANLİ*001
Record Dates: First submitted 2025-04-10; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Prenatal Attachment; Childbirth Preparation Program; Antenatal Education; Paternal Behavior
Keywords: Childbirth Preparation Program; Paternal attachment; Antenatal attachment; Midwifery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Father-Sensitive Birt Education (Experimental): The father-sensitive birth education group was given "Father-Sensitive Childbirth Preparation Education" consisting of four sessions.
  Interventions: Behavioral: Father-Sensitive Education
- Standardized Birt Education (Active Comparator): The control group received a total of 12 hours of standard childbirth preparation training, consisting of four three-hour sessions.
  Interventions: Behavioral: Standardized birth education

INTERVENTIONS:
Behavioral: Father-Sensitive Education — he father-sensitive education program preserves the basic structure of the Childbirth Preparation Education program, but has been enriched with original content that supports the active emotional and functional participation of fathers-to-be in the birth process.
  Arms: Father-Sensitive Birt Education
Behavioral: Standardized birth education — The control group received a total of 12 hours of standard childbirth preparation training, consisting of four three-hour sessions.
  Arms: Standardized Birt Education

SUMMARY:
This study was planned as a randomised controlled trial to examine the effects of a "Father-Sensitive Childbirth Preparation Class" on the level of prenatal attachment. The main question it aims to answer is:

1- How does a father-sensitive birth preparation class affect fathers' prenatal attachment levels?

It was conducted between February 1, 2024, and October 1, 2024, with expectant fathers living in Mersin province, whose spouses were experiencing their first pregnancy, who were between 20-32 weeks' gestation, and who were going to become fathers for the first time.

A total of 99 expectant fathers were included in the study - 50 in the intervention group and 49 in the control group. The intervention group was given a "Father-Sensitive Childbirth Preparation Training" consisting of four sessions, while the control group received a standard "Childbirth Preparation Training", also consisting of four sessions.

The "Descriptive Data Collection Tool" and the "Prenatal Father Attachment Scale" were used to collect the research data.

ELIGIBILITY:
Inclusion Criteria:

Participants were:

* Over 19 years of age,
* At least literate,
* Whose spouse was between 20 and 32 weeks pregnant,
* Whose spouse was primigravida,
* Whose spouse had a singleton pregnancy,
* With no prior experience of pregnancy, childbirth, or parenting,
* With no history of miscarriage, curettage, or perinatal loss,
* Whose spouse had no pregnancy-related complications or risk factors,
* Who had not previously attended any childbirth preparation training, pregnancy information classes, or parenting courses.

Exclusion Criteria:

Participants were excluded if they:

* Had a spouse whose pregnancy was outside the 20-32 week gestation range,
* Had a spouse with a multiple pregnancy,
* Had any pregnancy-related complications or risk factors (high risk),
* Had prior experience of pregnancy, birth, or parenting,
* Had experienced miscarriage, curettage, or perinatal loss,
* Had previously attended any childbirth preparation training, pregnancy information classes, or parenting courses.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 99 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Paternal Antenatal Attachment Scale (PAAS) total score mean | 14 days after completing the 12-hour father-sensitive childbirth preparation class
  It consists of 16 questions in a 5-point Likert format, designed to evaluate the feelings and thoughts of expectant fathers towards the developing baby in the womb, based on their emotions, thoughts, and experiences over the past two weeks.
  Nine items on the scale are reverse-scored, and the total score ranges from 16 to 80; higher scores indicate a stronger level of antenatal attachment.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)